CLINICAL TRIAL: NCT03990558
Title: Recovery of Consciousness Following Intracerebral Hemorrhage
Acronym: RECONFIG
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Pitié-Salpêtrière Hospital (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Jan Claassen, Professor of Neurology, Columbia University
Other Study IDs: AAAS3574; 1R01NS106014-01A1 (NIH)
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Intra Cerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Primary ICH: Subject with acute brain injury will have data collected, including EEG, behavioral, clinical, and outcome measures.

SUMMARY:
The objectives of the RECONFIG clinical study are to :

1. To identify the time to the first diagnosis of cognitive motor dissociation (CMD) in intracerebral hemorrhage (ICH) patients and to investigate whether these patients will clinically follow commands earlier after the hemorrhage.
2. To determine whether CMD independently predicts long term functional outcomes (6-month mRS scores) in ICH patients, and is associated with long term cognitive and quality of life outcomes.
3. To determine the EEG response to verbal commands of the motor imagery paradigm between patients with and without sensory aphasia.

The overall goal is to determine predictors and the trajectory of neurological recovery.

DETAILED DESCRIPTION:
Unconsciousness is common after an acute brain injury such as a brain hemorrhage, and recovery is poorly understood. This lack of knowledge is a key impediment to the development of novel strategies to improve outcomes and is one of the main reasons that prognostication of recovery of consciousness and functional outcomes is inaccurate. One-fifth of clinically unconscious patients with acute brain injury are able to follow commands using a simple, bedside EEG motor imagery test that directly measures brain activity associated with the attempt to move. This state is called cognitive motor dissociation (CMD). Pilot data indicate that CMD patients are more likely to clinically recover consciousness and have better longterm functional outcomes than non-CMD patients. To integrate these findings into clinical practice, there is a need to better understand the trajectory of CMD. This will only be possible in a tightly-controlled study with a homogenous patient cohort that is well characterized early after the injury and captures long-term outcomes.

RECONFIG is a multicenter, prospective, cross-sectional observational study in patients who have a clinical diagnosis of intracerebral hemorrhage and that are unresponsive at the time of enrollment. One hundred and fifty subjects will be recruited over 4 years at 2 sites. Subjects will be assessed with behavioral measures and MRI during the acute hospitalization. Patients will be followed for 6 months to determine the functional outcome (primary outcome measure). Additionally, the investigator will study conscious intracerebral hemorrhage patients with intracerebral hemorrhage and aphasia to determine the impact of aphasia.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Diagnosis of primary ICH (i.e., related to hypertension or anticoagulants) on Head CT and/or MRI in the frontal lobe, thalamus, or striatocapsular region.
* Unresponsive to commands within 48 hours after onset of the bleed.
* English, Spanish or, French as the primary language.

Exclusion Criteria:

* Major bleeding in the cortex outside of the frontal lobe, cerebellum, or brainstem (judged as a cause for unconsciousness as per the attending neurointensivist).
* Other causes of ICH or different types of acute brain injury (e.g., traumatic brain injury).
* Severe cardiorespiratory compromise and similar acutely life-threatening conditions at the time of enrollment.
* Evidence of pre-morbid aphasia or deafness.
* Unconscious prior to ICH.
* Pregnancy.
* Prisoners.
* Health care proxy decides against study participation or decided for withdrawal of life sustaining therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unresponsive and responsive patients diagnosed with ICH.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Time to clinical command following | Hospital discharge (approximately 3 weeks)
  To investigate whether patients will clinically follow commands earlier after the hemorrhage.
Modified Rankin Scale (mRS) Score | 6 months
  A standardized interview that measures the degree of disability or dependence in the daily activities of people who have suffered causes of neurological disability. The mRS ranges from 0 to 6, with higher scores indicating worse outcome.

SECONDARY OUTCOMES:
Quality of Life in Neurological Disorders (Neuro-QoL T-score) | 6 months
  Neuro-QoL is a measurement system that evaluates and monitors the physical, mental, and social effects experienced by adults and children living with neurological conditions. The T-score is the standardized score with a mean of 50 and a standard deviation of 10.
  For Neuro-QoL measures, higher scores equal more of the concept being measured (e.g., more Fatigue, more Lower Extremity Function - Mobility). Thus, a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
Difference in EEG response rate to verbal commands of the motor imagery paradigm. | 6 months
  EEG response will be compared between patients with and without sensory aphasia.
Modified Telephone Interview for Cognitive Status (TICS) score | 6 months
  A standardized test of cognitive functioning that was developed for use in situations where in-person cognitive screening is impractical or inefficient. The 11 test items usually take less than 10 minutes to administer and score. All examinee responses are recorded verbatim. The individual item scores are summed to obtain the TICS Total score. The TICS Total score can be interpreted by means of four qualitative impairment ranges: Unimpaired, Ambiguous, Mildly Impaired, and Moderately to Severely Impaired.
  TICS Total score provides a measure of global cognitive functioning and can be used to monitor changes in cognitive functioning over time. Higher score represents less cognitive impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Claassen, MD, Principal Investigator — Associate Professor of Neurology
Locations (2):
- United States (2):
  - University of Miami and Jackson Health System (UM/JHS), Miami, Florida
  - Columbia University Medical Center, New York, New York